CLINICAL TRIAL: NCT06062966
Title: The Effects of IL-1 Blockade on Inotrope Sensitivity in Patients With Heart Failure (AID-HEART)
Acronym: AID-HEART
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20027160
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure
Keywords: Inotrope sensitivity; IL-1 Blockade; Subcutaneous (SC); Hepatitis B Virus (HBV); Hepatitis C Virus (HCV; 6 Minute Walk Test (6MWT)
MeSH Terms: conditions — Heart Failure; Hepatitis B; Hepatitis C | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: This is a pilot study designed to treat 20 subjects to provide the preliminary data necessary to inform the design of subsequent hypothesis-driven studies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — Anakinra 100 mg SC daily will be administered to sujects on chronic inotrope treatment who are not candidates for transplantation or left ventricular assist device (LVAD).

SUMMARY:
End-stage heart failure (HF) is a progressive illness with a mortality rate similar to most advanced cancers.Roughly 5% of patients with HF have end-stage disease that is refractory to medical therapy (stage D heart failure). When patients reach this point in their disease, the only treatments known to prolong life are cardiac transplantation or left ventricular assist devices. In patients who do not qualify for these options, or elect a palliative approach, inotropes are frequently used to improve hemodynamics through an increase in cardiac output and reduction in filling pressures. While inotropes provide profound symptomatic relief, these benefits are accompanied by significant risks of progressive adverse cardiac remodeling, arrhythmias, and sudden death. There is, therefore, an urgent need to develop strategies to reduce the dose or duration of inotrope use in the management of patients with stage D of HF.

DETAILED DESCRIPTION:
Heart failure (HF) represents a leading cause of morbidity and mortality worldwide. Despite improvements in treatments and widespread efforts to implement guideline directed medical therapies, a growing population of patients with end-stage HF has limited treatment options to improve their quality and quantity of life. When patients reach this point in their disease, the only treatments known to prolong life are cardiac transplantation or left ventricular assist devices. In patients who do not qualify for these options, intravenous (IV) drugs that directly stimulate increased cardiac output ("inotropes") are frequently used to offer symptomatic relief. Inotropes exert their pharmacologic effects through direct activation of the beta-adrenergic receptors in the heart that increase heart rate and contractility. Unfortunately, however, the relief of symptoms from inotropes is accompanied by dose-dependent increased risks of progressive adverse cardiac remodeling, arrhythmias, and sudden death. There is therefore an urgent need to develop treatments that minimize the dosing requirements for inotropes or improve responsiveness to these agents.

Inflammation has been recognized as a major pathophysiological contributor to HF. Interleukin (IL)-1 is a potent apical inflammatory cytokine that is abundant in HF patients and correlates with disease severity. Preclinical data have shown that IL-1 is sufficient to induce cardiac dysfunction, desensitize beta-adrenergic receptors (impaired responsiveness to inotropes), and reduce exercise capacity. Among the observed effects of IL-1 in these models of HF, the impaired responsiveness to inotropes showed the greatest signal-to-noise ratio, suggesting a large potential effect size for IL-1 blockade to translated to human subjects. In a 12-week pilot clinical trial in stable HF patients not receiving IV inotropes, daily administration of an IL-1 antagonist (anakinra) improved exercise capacity. However, IL-1 blockade has not yet been evaluated in patients with more advanced HF requiring inotrope therapy.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis for the clinic visit is stage D heart failure being on chronic stable dose of inotrope therapy (dobutamine or milrinone for the previous 28 days)
* Prior documentation of impaired left ventricular systolic function (ejection fraction <50%) at most recent assessment by any imaging modality (within 12 months)
* Stable dose of inotrope treatment without a recent hospitalization within the previous month
* Age ≥21 years and willing/able to provide written informed consent
* The patient is willing and able to comply with the protocol (i.e. self administration of the treatment, and exercise protocol).
* Screening plasma C-reactive protein levels >2 mg/L

Exclusion Criteria:

* Concomitant clinically significant comorbidities including (but not limited to) acute coronary syndromes, uncontrolled hypertension or orthostatic hypotension, tachy- or brady-arrhythmias, acute or chronic pulmonary disease or neuromuscular disorders affecting respiration that would interfere with the execution, interpretation, or completion of the study
* Recent (previous 3 months) or planned resynchronization therapy (CRT), or valve surgeries
* Previous or planned implantation of left ventricular assist devices or heart transplant within the next 3 months
* Recent (<14 days) use of immunosuppressive or anti-inflammatory drugs (including oral corticosteroids at a dose of prednisone equivalent of 0.5 mg/kg/day but not including inhaled or low dose oral corticosteroids or non-steroidal anti-inflammatory drugs)
* Chronic inflammatory disorder (including but not limited to rheumatoid arthritis, systemic lupus erythematosus)
* Active infection (of any type), including chronic/recurrent infectious disease (including HBV, HCV, and HIV/AIDS) - but excluding HCV+ with undetectable plasma RNA
* Prior (within the past 5 years) or current malignancy on targeted treatment - excluding carcinoma in situ [any location] or localized non-melanoma skin cancer
* Stage V kidney disease or on renal-replacement therapy
* Neutropenia (<1,500/mm3 or <1,000/mm3 in African-American patients)
* Pregnancy or breastfeeding
* Angina, hypertension, arrhythmias, electrocardiograph (ECG) changes, or other non-cardiac limitations that limit 6MWD obtained during the baseline testing
* Hypersensitivity to anakinra or to E. coli derived products

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percent reduction in high-sensitive C-Reactive Protein (hsCRP, a biomarker for IL-1 activity) | Months 1 and 3 of treatment
  Percent reduction in hsCRP (a biomarker for IL-1 activity) at 1 month and 3 months of anakinra treatment.

SECONDARY OUTCOMES:
Change of inotrope dose (over 24 hrs) as a percentage of baseline inotrope dose (over 24 hrs) | Months 1 and 3 of treatment
  Inotrope use increases the risk of morbidity and mortality in patients with stage D HF. We hypothesize that anti-inflammatory treatment with IL-1 blockade (anakinra) will improve sensitivity to inotropes and therefore reduce the dose of inotropes required to alleviate HF symptoms in patients with end stage HF.
Change in exercise capacity will be measured with a 6-minute walk test (6MWT) | Baseline, Months 1 and 3 of treatment
  The 6-minute walk test (6MWT) is strongly correlated with cardiac output and disease severity and is an independent predictor of HF hospitalizations and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Azita Talasaz, Principal Investigator — Virginia Coomonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States